CLINICAL TRIAL: NCT02857296
Title: Evaluative Research in the Process of Implementation of an Alternative Device to Hospitalization for People Homeless With Severe Psychiatric Disorders
Acronym: REDAP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_3681 - 5325
Record Dates: First submitted 2016-07-29; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-07

CONDITIONS: Severe Psychiatric Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Interviews as Topic; Observation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: interview and observation

SUMMARY:
The research project aims to analyze the implementation of a new health care system - "alternative device to hospitalization and crisis home for people without home" - whose objective is to provide the homeless and suffering from severe psychiatric disorders adequate care to prevent situations from seeking care or complication of their disease. This device, if it has the administrative and legal structure of the Twin Stop Health Care (LHSS), is based on the original concept of "Soteria House." This will build tools for evaluating the performance of care device by a process evaluation describing and analyzing what activity involves the device, This research seeks to analyze the experimental device in the early stages of its implementation. The observation and analysis of the program period will adjust the management arrangements of the device. The data and conclusions from this research will identify the contributions and benefits of such a device and analyze the difficulties encountered in its implementation.

ELIGIBILITY:
Inclusion Criteria:

Adults without home with severe psychiatric disorders utilizing the structure, adults who master the French language

Exclusion Criteria:

adults not mastered the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults without home, with severe psychiatric disorders;
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
socio-anthropological survey | 1 year
  Biographical interviews and three du'entretiens targeted series on the course therapy will be conducted

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille